CLINICAL TRIAL: NCT05831761
Title: Effectivness of Tramadol or Topic Lidocaine on Postoperative Analgesia in Laparoscopic Colorectal Resection.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Alenka Spindler-Vesel, asoc. prof., University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 151/03/09
Record Dates: First submitted 2021-01-20; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2021-03

CONDITIONS: Postoperative Pain
Keywords: postoperative analgesia; neuropathic pain; laparoscopic colorectal surgery
MeSH Terms: conditions — Pain, Postoperative; Neuralgia | interventions — Dipyrone; Passive Cutaneous Anaphylaxis; Lidocaine

STUDY DESIGN:
Intervention Model Description: 4 parallel groups with different method of analgesia after laparoscopic colorectal resection.
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomised by random number generator after meeting the inclusion criteria.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PCA (Experimental): Postoperative intravenous infusion of piritramid patient controlled analgesia (PCA) (piritramide 0.5 mg/ml; infusion 1,5 mg/h, bolus 1,5 mg, lock out 30 minutes)
  Interventions: Drug: Comparison of analgesic efficacy protocol
- PCEA (Experimental): Postoperative patient controlled epidural analgesia (epidural cathterer inserted into Th7-8 intervertebral space, 200 ml of 0.125% levobupivacaine, 4 mg of morphine, 0.075 mg of clonidine; infusion 5 ml/h, bolus 5 ml, lock out 30 minutes).
  Interventions: Drug: Comparison of analgesic efficacy protocol
- tramadol (Experimental): Continous postoperative infusion of tramadol 300 mg and metamizole 2,5 g (in 500 ml 0.9% NaCl, rate of infusion 40 ml/h)
  Interventions: Drug: Comparison of analgesic efficacy protocol
- lidocaine (Experimental): Postoperative topical lidocaine and PCA (piritramide 0.5 mg/ml; infusion 0.5 mg/h, bolus 1.5 mg, lock out 20 minutes)
  Interventions: Drug: Comparison of analgesic efficacy protocol

INTERVENTIONS:
Drug: Comparison of analgesic efficacy protocol — Comparison of 4 possible analgesic protocols
  Other Names: PCA priritramide; PCEA; tramadole and metamizole; PCA and topical lidocaine

SUMMARY:
Comparison of different postoperative analgesia after laparoscopic colorectal surgery

DETAILED DESCRIPTION:
Postoperative pain treatment should be multimodal and opioid sparing. Thoracic epidural analgesia could relieve pain after laparoscopic surgery. Although ERAS guidelines suggest to use less invasive pain relieve technique, opioids are widely used perioperatively, despite of their side effects. Non-opioids and 5% lidocaine patches, used topicaly, could effectively reduce opioid consumption and their side effects.

Namely, efficient perioperative pain treatment is important to prevent late neuropathic pain, also after laparoscopic lower abdominal surgery. Its incidence is usually low compared to open surgery.

The aim of present study was to evaluate, if opioid consumption in laparoscopic colorectal surgery could be reduced with lidocaine patch at the wound site or with infusion of metamizole and tramadol and if the results meets epidural analgesia. We also compared the incidence of postoperative neuropathic pain among groups.

Prospective, randomised trial with 4 parallel groups was conducted at the University medical centre (UMC) Ljubljana. ASA (American Society of Anaesthesiologists) Class 2-3 high risk surgical patients from the Clinical department of abdominal surgery were included in the study. Adult patients that underwent laparoscopic colorectal surgery were included.

ELIGIBILITY:
Inclusion Criteria:

* scheduled elective laparoscopic colorectal surgery

Exclusion Criteria:

* critical preoperative state, pregnant women, laparotomy and palliative procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2009-09-01 (Actual); Primary Completion 2011-10-01 (Actual); Study Completion 2013-10-01 (Actual)

PRIMARY OUTCOMES:
Total opioid consumption | 0-48 hours after surgical procedure
  Measurement of piritramide consumprion
Presence of neuropathic pain | first 3 months after surgery
  Detecting of neuropathic pain using DN4 and PainDetect Questionnaire. These are clinically validated tools for detecting the presence of neuropathic pain and evaluating the severity.

CONTACTS AND LOCATIONS:
Overall Officials: Matej Jenko, Principal Investigator — University Medical Centre Ljubljana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kaba A, Laurent SR, Detroz BJ, Sessler DI, Durieux ME, Lamy ML, Joris JL. Intravenous lidocaine infusion facilitates acute rehabilitation after laparoscopic colectomy. Anesthesiology. 2007 Jan;106(1):11-8; discussion 5-6. doi: 10.1097/00000542-200701000-00007. PMID 17197840
- [Result] Tikuisis R, Miliauskas P, Samalavicius NE, Zurauskas A, Samalavicius R, Zabulis V. Intravenous lidocaine for post-operative pain relief after hand-assisted laparoscopic colon surgery: a randomized, placebo-controlled clinical trial. Tech Coloproctol. 2014 Apr;18(4):373-80. doi: 10.1007/s10151-013-1065-0. Epub 2013 Sep 13. PMID 24030782